CLINICAL TRIAL: NCT00559364
Title: A Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled, Phase III Study to Assess the Safety and Efficacy of Viokase® 16 for the Correction of Steatorrhea in Patients With Exocrine Pancreatic Insufficiency
Brief Title: Safety and Efficacy Study of Viokase® 16 for the Correction of Steatorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIO16EPI07-01
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Exocrine Pancreatic Insufficiency; Chronic Pancreatitis; Pancreatectomy
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis, Chronic | interventions — Proton Pump Inhibitors; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viokase® 16 (Experimental)
  Interventions: Drug: Viokase® 16; Drug: Proton pump inhibitor (PPI); Drug: Omeprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Proton pump inhibitor (PPI); Drug: Omeprazole

INTERVENTIONS:
Drug: Viokase® 16 — Patients assigned to Viokase® 16 will be given 22 tablets orally daily (that is, 6 tablets per meal and 2 tablets with 2 of 3 snacks) for 6 to 7 days in treatment phase.
  Arms: Viokase® 16
Drug: Placebo — Patients assigned to placebo will be given 22 matching placebo tablets orally daily (that is, 6 tablets per meal and 2 tablets with 2 of 3 snacks) for 6 to 7 days in treatment phase.
  Arms: Placebo
Drug: Proton pump inhibitor (PPI) — Patients on PPI during Screening will continue their usual PPI therapy throughout the study.
Drug: Omeprazole — Patients not using PPI therapy at Screening will be given omeprazole 20 milligram orally once daily throughout the study.

SUMMARY:
This study assesses the efficacy and safety of Viokase® 16 for the correction of steatorrhea (malabsorption of dietary fats) in patients with a history of exocrine pancreatic insufficiency (EPI) due to chronic pancreatitis (CP) or pancreatectomy. This study is sponsored by Aptalis Pharma (formerly Axcan).

DETAILED DESCRIPTION:
This study is a Phase III, multicenter, randomized, double-blind, parallel, placebo-controlled study, to assess the efficacy and safety of Viokase® 16 for the correction of steatorrhea in patients with EPI due to CP or pancreatectomy. The study will include the following phases: screening phase (up to 10 days), wash-out phase (6 to 7 days), randomization phase (up to 10 days), and treatment phase (6 to 7 days).

In screening phase, patients will undergo screening procedures prior to entry into the study.

In wash-out phase, stool collection will be performed to allow determination of the baseline CFA.

In randomization phase, patients who qualify for the Treatment Phase (that is, patients who have a CFA% below 80%) will be randomized in the study.

In the treatment phase, patients will be randomized in a 2:1 ratio (Viokase® 16 or Placebo). In treatment phase, stool collection period will be performed to allow determination of the CFA% that will serve to assess the efficacy of Viokase® 16 for the correction of steatorrhea. Follow-up procedures will be scheduled 7 to 10 days after discharge. Patients who do not show abnormal findings, adverse events or concomitant medications during the treatment phase will be assessed via follow-up telephone call. Patients who show abnormal findings (physical examination, vital signs, clinical laboratory tests, adverse events, concomitant medications) during the treatment phase will complete a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be male or female, aged 18-80 years
* Patients must have the ability to provide informed consent
* Female patients of childbearing potential must have a negative pregnancy test at screening, must use adequate contraception prior to and during the study and must agree not to attempt to become pregnant during the study; and female patients of non-childbearing potential must be surgically sterile or postmenopausal for at least 12 consecutive months
* Patients must have a medical condition compatible with EPI such as chronic pancreatitis or partial or total resection of the pancreas
* Patients with CP due to alcohol abuse may be included provided they show no clinical symptoms of recent alcohol consumption and no alcohol withdrawal symptoms
* Patients with CP must have at least one of the following conditions: an abnormal secretin test, diffuse calcification of the pancreas on plain film of the abdomen, an abnormal endoscopic retrograde cholangiopancreatography (ERCP) or endoscopic ultrasound, an abnormal computed tomography (CT) (dilated main pancreatic duct, atrophy or calcification of the pancreas) or serum trypsin concentration below 20 nanogram per milliliter (ng/mL)
* Patients must have evidence of EPI as demonstrated by a fecal elastase (FE-1) determination equal to or below 100 microgram/gram (mcg/g) of stools (FE-1 ScheBo test) at screening
* Patients must have evidence of EPI as manifested by a CFA% below 80% after the wash-out phase
* Patients must be able to comply with a high-fat diet

Exclusion Criteria:

* Patients with a known hypersensitivity and/or contraindication to any of the study medications, to their excipients, components or to Federal Food, Drug, and Cosmetic (FD and C) Blue No. 2 dye marker
* Patients with acute pancreatitis or with an acute exacerbation of CP at screening or within the last 2 weeks before screening
* Patients with any active or recurrent malignant pancreatic tumor
* Patients with a history of significant bowel resection
* Patients with a dysmotility disorder
* Patients with insufficient body mass (body mass index less than 18)
* Patient not willing to be off therapeutic doses for at least 7 days prior to study entry and throughout the course of the study, medications or products that could interfere with fecal fat excretion
* Patients who do not limit alcohol intake to less than or equal to 1 drink per day during screening and randomization phases and patients who do not refrain from drinking during inpatient periods of the study
* Patients who have been treated with the following drugs within 7 days prior to screening: H2-receptor antagonists, gastrointestinal anticholinergics and antispasmodics
* Patients known to have a significant medical and/or mental disease that would compromise the patient's welfare or confound the study results
* Patients with a history of fibrosing colonopathy, cirrhosis of the liver, or portal hypertension
* Patients who have a condition known to increase fecal fat loss including celiac disease, biliary cancer, biliary stricture, cholelithiasis, Crohn's disease, pancreatic cancer, radiation enteritis, tropical sprue, whipple's disease, lactose intolerance, pseudomembranous colitis
* Female patients who are pregnant or breastfeeding
* Patients who have received an investigational drug within 30 days prior to entering the screening phase of the study
* Patients with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels greater than 3 times the upper limit of normal values or elevated uric acid levels greater than 1.5 times the upper limit of normal values
* Patients with causes for EPI other than CP and partial/total pancreas resection, example, cystic fibrosis, primary sclerosing cholangitis, hemochromatosis, isolated enzyme deficiency, deficiency in activation of enzymes in the small intestine etc
* Patients with a history or clinical evidence of any relevant cardio- or cerebrovascular, renal, endocrine, neurologic, infectious, other gastrointestinal, hematological, oncological or psychiatric disease or emotional problems, which, in the opinion of the investigator, would pose a significant risk for the patient, invalidate the giving of informed consent or limit the ability of the patients to comply with study requirements or interfere otherwise with the conduct of the study and the same applies for immunocompromised patients and/or neutropenic patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (18):
- Darmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States
- Hotel-Dieu de Levis, Lévis, Quebec, Canada
- Poland (12):
  - III Oddzial Chorób Wewnetrznych i Gastroenterologii, Bialystok
  - Akademickie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Centralny, Katowice
  - Klinika Chorob Wewnetrznych z Poliklinika, Krakow
  - Uniwersytecki Szpital Kliniczny nr 1 im, Lodz
  - SP Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Wojewodzki Szpital Specjalistyczny Nr5, Sosnowiec
  - SP Szpital Kliniczny nr 1 Klinika Gastroenterologii, Szczecin
  - Klinika Gastroenterologii i Chorób Przemiany Materii, Warsaw
  - Klinika Chorob Wewnetrznych i Gastroenterologii, Warsaw
  - Wojewodzki Szpital Brodnowski, Warsaw
  - Katedra Klinika Gastroenterologii, Wroclaw
- Slovakia (4):
  - University Hospital Brastislava, Brastislava
  - University Hospital Bratislava, Bratilslava
  - NZZ Management spol.S.r.o., Nitra
  - Gastro I. s.r.o., Gastroenterologicka, Prešov

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients underwent screening phase (up to 10 days) and wash-out phase (6 to 7 days, where baseline coefficient of fat absorption [CFA] was determined) before entering randomization phase. Out of 218 patients, who entered screening and washout phases, 168 discontinued due to screen failure; 50 patients were randomized to treatment phase.
Groups:
- Viokase®: Patients received Viokase® 16, 22 tablets orally daily (that is, 6 tablets per meal and 2 tablets with 2 of 3 snacks) for 6 to 7 days in treatment phase. Patients on proton pump inhibitor (PPI) therapy during Screening continued their usual (those not using PPI therapy at screening received omeprazole 20 milligram orally once daily) throughout the study.
- Placebo: Patients received matching placebo, 22 tablets orally daily (that is, 6 tablets per meal and 2 tablets with 2 of 3 snacks) for 6 to 7 days in treatment phase. Patients on proton pump inhibitor (PPI) therapy during Screening continued their usual (those not using PPI therapy at screening received omeprazole 20 milligram orally once daily) throughout the study.
Period: Overall Study
Arm/Group | Viokase® | Placebo
Started | 30 | 20
Completed | 29 | 20
Not Completed | 1 | 0
Not completed — Inclusion/exclusion criteria failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Viokase® | Placebo | Total
Number analyzed (Participants) | 30 | 20 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (9.91) | 50.6 (7.63) | 50.8 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percent Coefficient of Fat Absorption (CFA)
Description: Percent CFA was calculated as ([fat intake - fat excretion]/fat intake)*100, determined in the stools which was collected from Day 1 to Day 4 or Day 5 during the inpatient period of treatment phase. Mean percent (%) CFA was calculated for Day 1 to Day 4 or Day 5 in inpatient period of treatment phase.
Time Frame: Day 1 up to Day 4 or Day 5 in inpatient period of treatment phase
Population: Intent-to-treat (ITT) population included all randomized patients. Missing values at treatment phase were imputed using the median (50th percentile) of all non-missing values within a treatment group.
Measure: Mean (Standard Deviation); unit: percent CFA
Arm/Group | Viokase® | Placebo
Number analyzed (Participants) | 30 | 20
percent CFA | 85.52 (8.902) | 58.02 (24.249)
Statistical Analysis 1: Comparison: Viokase® vs Placebo; Analysis of covariance (ANCOVA) model using treatment group and pooled site as fixed effects and wash-out phase CFA% value as covariate was used; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Mean Daily Number of Stools
Description: Mean daily number of stools of each patient was calculated from frequency of stools by the patient per day. Mean daily number of stools during the collection period (Day 1 to Day 4 or Day 5 in inpatient period of treatment phase) for total patients was summarized.
Time Frame: Day 1 up to Day 4 or Day 5 in inpatient period of treatment phase
Population: ITT population included all randomized patients.
Measure: Mean (Standard Deviation); unit: stools per day
Arm/Group | Viokase® | Placebo
Number analyzed (Participants) | 30 | 20
stools per day | 1.93 (0.989) | 2.33 (0.950)

3. Secondary Outcome: Percentage of Stools Categorized as Per Consistency
Description: Stool consistency was categorized as hard, formed/normal, soft and watery. Percentage of stools of a specific consistency for each patient was calculated as: (total number of stools of specific consistency during the completed days of the inpatient period/ total number of stools during the completed days of the inpatient period)*100. Mean percentage of stool categorized as per consistency for total patients was summarized.
Time Frame: Day 1 up to Day 4 or Day 5 in inpatient period of treatment phase
Population: ITT population included all randomized patients.
Measure: Mean (Standard Deviation); unit: percentage of stools
Arm/Group | Viokase® | Placebo
Number analyzed (Participants) | 30 | 20
percentage of stools
  Hard stools | 5.08 (13.61) | 0.67 (2.98)
  Formed/normal stools | 45.86 (33.27) | 37.23 (37.91)
  Soft stools | 47.80 (33.31) | 55.48 (39.46)
  Watery stools | 1.26 (4.82) | 5.80 (14.57)

ADVERSE EVENTS:
Time Frame: Day 1 of treatment phase up to 30 days after last dose administration
Description: Adverse event (AE) was any untoward medical occurrence regardless of causal relationship to study drug. Serious AE was any event that resulted in death, life threatening, required or prolonged in-patient hospitalization, significant disability/incapacity, or was a congenital anomaly/birth defect or is assessed as important medical event.
Arm/Group | Viokase® | Placebo
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/20
Other Adverse Events (participants affected / at risk) | 7/30 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Viokase® (N=30) | Placebo (N=20)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Coagulation factor decreased (Investigations) | 1 | 0
Disease progression (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Viokase® (N=30) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anal pruritus (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Results for percentage of stool characteristics per bowel movement and number of days with at least 1 stool of specific characteristic were not reported due to change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions vary in accordance with each agreement with the individual investigators. Sponsor will allow publication but will prohibit disclosure of Sponsor's confidential information within any publication and can defer publication for a period of time to allow for Sponsor to obtain patent or other intellectual property right protection.